CLINICAL TRIAL: NCT01336816
Title: A Randomized, Double-Blinded, Placebo-Controlled, Crossover, Pilot Study to Evaluate the Efficacy of Ariva® Silver Wintergreen, a Smoking Aversive Lozenge, Containing Tobacco and Silver Salt - in Healthy Smokers
Brief Title: A Pilot Study to Evaluate the Efficacy of Ariva® Silver Wintergreen, a Smoking Aversive Lozenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Star Scientific, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: SSI-042
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Tobacco Use Disorder; Smoking
Keywords: smoking; smokeless; aversion; nicotine; nicotine replacement
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ariva Silver Wintergreen (Experimental): Subjects allow study product lozenge to dissolve in mouth, smoke a cigarette, then answer questionnaires about product taste and effect on desire to smoke.
  Interventions: Other: Ariva Silver Wintergreen
- Placebo Wintergreen (Placebo Comparator): Subjects allow study placebo lozenge to dissolve in mouth, smoke a cigarette, then answer questionnaires about product taste and effect on desire to smoke.
  Interventions: Other: Placebo Wintergreen

INTERVENTIONS:
Other: Ariva Silver Wintergreen — Study product containing 6 mg silver salt and 2 mg nicotine per dissolvable lozenge, administered orally as a single dose.
  Arms: Ariva Silver Wintergreen
Other: Placebo Wintergreen — Placebo Wintergreen lozenge containing no tobacco, nicotine, or silver salt, administered orally as a single dose.
  Arms: Placebo Wintergreen

SUMMARY:
This is a study to determine the safety and effectiveness of silver salt in Ariva® Silver Wintergreen Lozenge on discouraging smoking, by its imparting an unfavorable taste to the smoker when tobacco is smoked.

DETAILED DESCRIPTION:
Each subject will be given an Ariva® Silver Wintergreen lozenge or a Placebo Wintergreen lozenge on a random basis.

Once the lozenge has dissolved in the mouth, subjects will smoke one of their own cigarettes, and will answer questions about the experience and their craving for a cigarette.

After a washout period, each subject will repeat the steps with the second type of lozenge.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult smoker
* smoking for at least 5 years
* smoking at least one (1) pack of cigarettes a day
* interest in quitting smoking

Exclusion Criteria:

* known allergy to silver or silver salts
* pregnant or breast-feeding
* current drug or alcohol abuse, and/or history of drug or alcohol dependence within 3 months of study

Ages: 23 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Ariva® Silver Wintergreen lozenge on discouraging smoking in smokers | 90 minutes
  Effectiveness measured by change in scores over time across several questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Varga, MD, Principal Investigator — Star Scientific, Inc
Locations (1):
- Comfort Inn, Martinsburg, West Virginia, United States